CLINICAL TRIAL: NCT06128317
Title: Cardiac Biochemical and Omics-based Biomarkers in Patients Presenting Symptoms of Acute Coronary Syndrome in the Emergency Department (ACS Registry)
Brief Title: Myocardial Infarction Registry
Acronym: MIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mustafa Yildirim, Dr. med. univ., University Hospital Heidelberg
Other Study IDs: MIR
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine blood samples at presentation, a second blood sample for study purposes will be collected after 1 hour of the first index visit. On the routine follow-up visit, we will collect 20 ml for storage in addition to the routine blood test. Blood samples will be obtained by standard venous blood sampling. Assessment of parameters include laboratory values with special focus on findings related to myocardial injury as indicated by high sensitivity cardiac troponin T (hs-cTnT) and hs-cTnI. Moreover, the laboratory panel comprises other cardiac biomarkers, electrolytes, renal (creatine, glomerular filtration rate) and liver function (GOT, GPT, LDH), C-reactive protein, D-dimer etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIR (Myocardial Infarction Registry): All patients presenting to the Emergency Department with suspected acute coronary syndrome
  Interventions: Other: no intervention is intended.

INTERVENTIONS:
Other: no intervention is intended. — no intervention is intended.

SUMMARY:
The single-center MIR-registry was created to assess real-world prevalence, demographic characteristics and management of patients with acute coronary syndrome presenting in the emergency department (ED) of University of Heidelberg.

DETAILED DESCRIPTION:
To conduct a comprehensive characterization of patients with symptoms of acute coronary syndrome or elevated troponin levels. Records include clinical routine parameters, there will be an expansion involving the collection of blood samples for the analysis of novel laboratory-based and omics-based biomarkers. The ACS registry is monothetically managed by the Department of Internal Medicine III at Heidelberg University Hospital and is intended to serve as a basis for further clinical diagnostic and outcome studies. The blood samples will serve as the foundation for a comprehensive analysis of established and novel laboratory-based markers, as well as omics-based biomarkers (miRNA, metabolomics, and proteomics). Follow-up was performed via review of medical reports, phone calls and postal queries. The outcome parameters comprised rates for all-cause mortality, non-hemorrhagic stroke, myocardial infarction, and hospitalization for any cause.

ELIGIBILITY:
Inclusion Criteria:

The study will include consecutive patients who present to the cardiology emergency department at Heidelberg University Hospital with symptoms of acute coronary syndrome or a troponin increase (hs-TnT >14 ng/L). Additional inclusion criteria are a minimum age of 18 years and providing informed consent through written consent to participate in the study. The following medical conditions are intended to be distinguished from one another:

* Acute myocardial infarction
* Unstable angina pectoris
* Myocarditis
* Heart failure
* Cardiomyopathies
* Pulmonary embolism
* Renal insufficiency
* Supraventricular and ventricular tachycardias
* Hypertensive crisis
* Non-cardiac chest pain

Exclusion Criteria:

Exclusion criteria are defined according to GCP (Good Clinical Practice), i.e., mental illnesses/dementia (lack of capacity to provide informed consent), pregnancy/breastfeeding, as well as acute conditions requiring immediate treatment (e.g., cardiogenic shock).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort consisting of consecutive patients with suspected acute coronary syndrome presenting to the emergency department of the Heidelberg University Hospital.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 12 months
  all-cause mortality during follow-up

SECONDARY OUTCOMES:
myocardial infarction | 12 months
  myocardial infarction during follow-up
stroke | 12 months
  stroke during follow-up
Rehospitalization | 12 months
  Rehospitalization during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim M, Salbach C, Mueller-Hennessen M, Frey N, Giannitsis E. Comparative Analysis of Single- and Dual-Marker Strategies for Rapid Non-ST-Segment-Elevation Myocardial Infarction Rule-Out Using Cardiac Myosin-Binding Protein C, Copeptin, and High-Sensitivity Cardiac Troponin T in the Emergency Department. J Am Heart Assoc. 2025 May 20;14(10):e039379. doi: 10.1161/JAHA.124.039379. Epub 2025 May 13. PMID 40357668